CLINICAL TRIAL: NCT01683175
Title: A Prospective, Open-labelled, Randomized, Multicenter Phase II Study to Evaluate Efficacy and Safety of Erlotinib vs NP Chemotherapy as Adjuvant Therapy in Post Radical Operation NSCLC Patients With EGFR19 or 21 Exon Mutation
Brief Title: Erlotinib in Post Radical Operation NSCLC Patients With EGFR Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28280
Record Dates: First submitted 2012-08-30; First posted 2012-09-11 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Non-small Cell Lung Cancer Stage III
Keywords: Erlotinib; adjuvant therapy; radical operation; IIIA NSCLC; EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Cisplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Erlotinib 150mg daily oral up to 2 years
  Interventions: Drug: Erlotinib
- Arm 2 (Active Comparator): NP Chemotherapy for 4 cycles
  Interventions: Drug: cis-platinum; Drug: Vinorelbine

INTERVENTIONS:
Drug: Erlotinib
  Arms: Arm 1
Drug: cis-platinum
  Arms: Arm 2
Drug: Vinorelbine
  Arms: Arm 2

SUMMARY:
This study is to compare 2-year Disease Free Survival Rate (DFSR) in post radical operation IIIA Non-Small Cell Lung Cancer (NSCLC) patients with Epidermal Growth Factor Receptor (EGFR) 19 or 21 exon mutation treated Erlotinib vs NP chemotherapy as adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* IIIA NSCLC patients according to TMN-staging of Lung Staging Standard version 7 2009, confirmed by histopathology or cytology after radical operation, and having EGFR exon 19 deletion mutation or exon 21 L858R single base substitution;
* Accept study adjuvant therapy within 6 weeks post radical operation;
* ECOP PS 0-1; Life expectancy ≥12 weeks;
* Hematology: absolute neutrophil count (ANC) ≥1.5×10^9/L; platelet count ≥100×10^9/L; hemoglobin concentration ≥ 9.0 g/dL (permit to maintain hematologic criteria by blood transfusion);
* Liver Function: TBil ≤1.5xULN; ALT and AST ≤2.5xULN;
* Renal Function: Cr ≤1.25xULN, and Ccr ≥60ml/min;
* Female patients of childbearing potential must have a negative serum or urine pregnancy test within 7 days before study treatment;
* Signed inform consent form by patient or his/her legal representative;
* Comply with study protocol and procedure, and be able to take oral medication; Aged ≥18 years and ≦75 years;
* Eligible patients of reproductive potential (both sexes) must agree to use a reliable method of birth control before enrollment, during the study period and for at least 30 days after their last dose of study therapy;

Exclusion Criteria:

* Having treated by Her-Target therapy, i.e. erlotinib, gefitinib, cetuximab, trastuzumab;
* Having treated by any systemic anti-tumor therapy of NSCLC, including cytotoxic therapy, target medication treatment (i.e. monoclonal antibody), investigational therapy;
* Having local radiotherapy of NSCLC; Upper gastrointestinal physiological disorders, or malabsorption syndrome, or intolerance of oral medication, or active peptic ulcer;
* The findings in radical operation are lymph nodes with extracapsular invasion, or fusion, or all of dissection lymph nodes positive by pathology;
* Diagnosed other malignant tumor besides NSCLC within 5 years prior the study treatment (except having simple surgical resection with 5-year disease free survival,cured in situ of cervical carcinoma, cured basal cell carcinoma and bladder epithelial tumor);
* Confirmed recurrent cancer by Clinical objective evidence (pathology or radiography images) before the study adjuvant therapy;
* Known hypersensitivity to platinum, Vinorelbine, EGFR-TKI agents or relevant components in the formulation;
* Uncontrolled eye inflammation or infection, or any potential circumstances lead to eye inflammation or infection;
* Active interstitial lung disease (ILD) by any clinical evidence; patients with any co-morbidities, or motalic disorders, or any abnormal findings in physical examination or laboratory tests are suspected to have contraindication of study therapy or high risk of study treatment complications;
* Any unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, angina starting in latest 3 months, Congestive heart failure (NYHA ≥ II), myocardial infarction within 6 months prior enrollment, under medication treatment of severe arrhythmia, liver, renal or metabolic disease;
* know HIV infection Pregnant or breastfeeding women;
* ECOG PS ≥2;
* Mixed with small cell lung cancer;
* Other conditions investigators evaluate that patient is not eligible to this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-08; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
2-year disease free survival rate (DFSR) | 2 years
  2-year disease free survival rate is defined as the estimation percentage of disease free survival patients with study treatment at 2-year.

SECONDARY OUTCOMES:
disease free survival | 5 years
  Disease free survival is defined as the time from randomization to disease recurrence or death which comes first.
overall survival (OS) | 5 years
  Overall survival is defined as the time from randomization to death.
Quality of Life | 5 years
  The score of Functional Assessment of Cancer Therapy - Lung (FACT-L) subscale and Lung Cancer Symptom Scale (LCSS)
Adverse Event (AE) | 5 years
  frequency of Adverse Event
Serious Adverse Event (SAE) | 5 years
  Frequency of Serious Adverse Event (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Changli Wang, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (15):
- China (15):
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Beijing Cancer Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The second people's hospital of Sichuan, Chengdu
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The third affiliated hospital of Harbin Medical Univer, Harbin
  - The affiliated hospital of medical college Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Hebei Provincial Tumor Hospital, Shijiazhuang
  - The first affiliated hospital of Soochow University, Suzhou
  - The fourth military medical university，Tangdu Hospital, Xi'an

REFERENCES:
- [Derived] Occhipinti M, Imbimbo M, Ferrara R, Simeon V, Fiscon G, Marchal C, Skoetz N, Viscardi G. Adjuvant epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKIs) for the treatment of people with resected stage I to III non-small-cell lung cancer and EGFR mutation. Cochrane Database Syst Rev. 2025 May 27;5(5):CD015140. doi: 10.1002/14651858.CD015140.pub2. PMID 40421698
- [Derived] Yue D, Xu S, Wang Q, Li X, Shen Y, Zhao H, Chen C, Mao W, Liu W, Liu J, Zhang L, Ma H, Li Q, Yang Y, Liu Y, Chen H, Zhang Z, Zhang B, Wang C. Updated Overall Survival and Exploratory Analysis From Randomized, Phase II EVAN Study of Erlotinib Versus Vinorelbine Plus Cisplatin Adjuvant Therapy in Stage IIIA Epidermal Growth Factor Receptor+ Non-Small-Cell Lung Cancer. J Clin Oncol. 2022 Dec 1;40(34):3912-3917. doi: 10.1200/JCO.22.00428. Epub 2022 Aug 26. PMID 36027483
- [Derived] Yue D, Xu S, Wang Q, Li X, Shen Y, Zhao H, Chen C, Mao W, Liu W, Liu J, Zhang L, Ma H, Li Q, Yang Y, Liu Y, Chen H, Wang C. Erlotinib versus vinorelbine plus cisplatin as adjuvant therapy in Chinese patients with stage IIIA EGFR mutation-positive non-small-cell lung cancer (EVAN): a randomised, open-label, phase 2 trial. Lancet Respir Med. 2018 Nov;6(11):863-873. doi: 10.1016/S2213-2600(18)30277-7. Epub 2018 Aug 24. PMID 30150014